CLINICAL TRIAL: NCT04812665
Title: Feasibility Study of Digital Health for Caregivers Emotional and Self-management Support of Children Receiving Growth Hormone Treatment
Brief Title: Digital Health for Caregivers Emotional and Self-management Support
Acronym: CARING
Status: Completed | Type: Observational
Sponsor: Adhera Health, Inc. (Industry)
Collaborators: Hospital Miguel Servet (Other); Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: CAR-0220
Record Dates: First submitted 2021-03-17; First posted 2021-03-24 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Emotional Adjustment; Mood Disturbance
Keywords: Emotional Adjustment; Mood Disturbance; Behavioral Intervention; mHealth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Qualitative sub-study (SS1): One group of caregivers (n = 10) will engage with the mHealth solution during 1 month. Subsequently, an individual semi-structured interview with each of the participants will proceed to gather user experience qualitative information.
  Interventions: Behavioral: mHealth solution based on emotional and behavioral change techniques
- Quantitative sub-study (SS2): A different group of caregivers (n = 55) will engage with the mHealth solution during 3 months. As elaborated in the following sections, a quantitative approach will be adopted to assess different emotional, behavioral and growth parameters before and after engaging with the mHealth solution (pre-post design).
  Interventions: Behavioral: mHealth solution based on emotional and behavioral change techniques

INTERVENTIONS:
Behavioral: mHealth solution based on emotional and behavioral change techniques — Adhera supports the empowerment of patients with chronic conditions by supporting the acquisition of healthier lifestyles, improved mental wellbeing and grounded on the principles of behavioral change.
  The solution is based on incorporating the principles of personalized health education into a mobile platform which is achieved by applying the Integrated Model of Behavioral Change which is further adapted using recommender systems. Emotional and mental health elements, such as stress, resilience, are crucial part in the acquisition of self-management behaviors and will be the main focus of this intervention. Adhera adapts to provide tailored support to specific users' needs.
  Other Names: Adhera

SUMMARY:
This feasibility study builds upon mental health and technology acceptance theoretical frameworks. It seeks to examine potentials of a novel mobile Health (mHealth) solution based on emotional and behavioral change techniques, to provide emotional and self-management tailored support to caregivers of children undergoing Growth Hormone treatment (GHt).

DETAILED DESCRIPTION:
This feasibility study builds upon mental health and technology acceptance theoretical frameworks. It seeks to examine potentials of a novel mobile Health (mHealth) solution based on emotional and behavioral change techniques, to provide emotional and self-management tailored support to caregivers of children undergoing Growth Hormone treatment (GHt).

Primary Objectives:

* To gather qualitative information enabling to better understand individualized experiences of caregiving children undergoing GHt and perceived barriers/facilitators for adoption of the mHealth solution.
* To assess positive mood states of caregivers of GHt patients as an indicator of emotional wellbeing related to the use of the mHealth solution.

Secondary Objectives:

To explore whether the mHealth solution applied to caregivers of children undergoing GHt might affect:

* Broader emotion-related parameters: Distress (emotional disturbance), self-efficacy (perceived own capability of managing stress), and general psychological wellbeing of caregivers.
* Perceived Health-related quality of life (HRQoL) of children (evaluated from the caregivers' perspective).
* Behavioral parameters: Usability / engagement with the mHealth solution and children's adherence to treatment measured by Easypod-Connect.
* Growth parameters: height of the child.

ELIGIBILITY:
The study targets caregivers of GHt patients.

Inclusion Criteria:

* Adherence to GHt monitored in the last month prior enrollment indicates a ratio less than 85%.
* Legal guardian of children who receive GHt in accordance with approved indications in Spain.
* Explicit agreement on data sharing regarding adherence to GHt gathered through the Easypod Connect.
* Participants must be able to interact with a smart phone and willing to install the mHealth solution of the study in their smart phone.
* Participants must sign the specific informed consent form for the study.

Exclusion Criteria:

* Candidates without an smart phone or not being able to interact with it.
* Only one legal guardian per child can participate in the study.
* Participants of SS1 will not take part in SS2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample of the study (caregivers) will be recruited from the Pediatric Endocrinology unit at the Miguel Servet Children's University Hospital. This public hospital provides pediatric healthcare delivery to the regional area of Zaragoza (Spain), which covers a total of 367.110 inhabitants.
  Participants will sign an informed consent during routine clinical visits to the centers. For accessing treatment adherence data (Easypod-Connect) of children aged 12 y.o. and over, a specific Informed Consent Form (ICF) will also need to be signed by the minor according to the Spanish regulation, jointly with the legal guardian's one.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Sub-study 1: Psychological burdens experienced as caregivers of children receiving GHt and barriers/facilitators for adopting the mHealth solution | 1 Month
  A semi-structured interview based on a mental health and technology acceptance theoretical framework has been specifically designed for this purpose
Sub-study 2: Changes on caregiver's positive mood | 3 Months
  Positive subscale of the Positive and Negative Affect Scale (PANAS). Scores can range from 10-50 for both the Positive and Negative Affect with the lower scores representing lower levels of Positive/Negative Affect and higher scores representing higher levels of Positive/Negative Affect.

SECONDARY OUTCOMES:
Emotional outcome: Changes on caregiver's distress | 3 Months
  Distress assessed with the depression, anxiety, and stress scale (DASS-21). DASS-21 is a self-report questionnaire consisting of 21 items, 7 items per subscale: depression, anxiety and stress. Patients are asked to score every item on a scale from 0 (did not apply to me at all) to 3 (applied to me very much). Sum scores are computed by adding up the scores on the items per (sub)scale and multiplying them by a factor 2. Sum scores for the total DASS-total scale thus range between 0 and 120, and those for each of the subscales may range between 0 and 42. Cut-off scores of 60 and 21 are used for the total DASS score and for the subscales respectively. Scores ≥60 (for DASS-total) and ≥21 (for the depression subscale) are labeled as "high" or "severe".
Emotional outcome: Changes on caregiver's general wellbeing | 3 Months
  Assessed with the short form of the Mental Health Continuum - short form questionnaire (MHC-SF). Total sum scores on the MHC-SF can range from 0 to 70, with higher scores indicating higher levels of well-being.
Emotional outcome: Changes on caregiver's perceived self-efficacy | 3 Months
  Perceived self-efficacy assessment with the General Self-Efficacy Scale (GSE), the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Health-related Quality of Life (HrQoL): Changes on child's HRQoL | 3 Months
  Children HRQoL assessment with KIDSCREEN-10 index answered by the caregiver as a proxy. The scores ranges between 10 and 50, and are linearly converted into 0-100 scale in which higher scores represent better quality of life.
Health-related Quality of Life (HrQoL): Changes on child's HRQoL | 3 Months
  Child HRQoL assessment with Quality of Life in Short Statured Youth (QoLISSY) questionnaire answered by the caregiver as a proxy. This version has 47 items with a 5-point likert scale each. Total score is linearly transformed into 0 to 100 scores with higher values representing higher HRQOL.
Behavioral outcome: Usability | 3 Months
  mHealth solution usability assessed with the System Usability Scale (SUS) questionnaire. SUS can range between 0 and 100 scores, with higher values representing higher usability.
Behavioral outcome: Treatment adherence | 3 Months
  Adherence to the Growth Hormone treatment (GHt) will be measured with the data collected by the Easypod Connect device.
Growth parameter: height | 6 Months
  Height is a crucial indicator of the growth of children under Growth Hormone therapy. Measures from 6 month before starting the study to the end of the study will be obtained from Patient's Electronic Health Record.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Fernández-Luque, PhD, Principal Investigator — Adhera Health, Inc.
Locations (1):
- Hospital Universitario Miguel Servet, Zaragoza, Aragon, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carrasco-Hernandez L, Jodar-Sanchez F, Nunez-Benjumea F, Moreno Conde J, Mesa Gonzalez M, Civit-Balcells A, Hors-Fraile S, Parra-Calderon CL, Bamidis PD, Ortega-Ruiz F. A Mobile Health Solution Complementing Psychopharmacology-Supported Smoking Cessation: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Apr 27;8(4):e17530. doi: 10.2196/17530. PMID 32338624
- [Background] Hors-Fraile S, Malwade S, Spachos D, Fernandez-Luque L, Su CT, Jeng WL, Syed-Abdul S, Bamidis P, Li YJ. A recommender system to quit smoking with mobile motivational messages: study protocol for a randomized controlled trial. Trials. 2018 Nov 9;19(1):618. doi: 10.1186/s13063-018-3000-1. PMID 30413176
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Mohr DC, Schueller SM, Montague E, Burns MN, Rashidi P. The behavioral intervention technology model: an integrated conceptual and technological framework for eHealth and mHealth interventions. J Med Internet Res. 2014 Jun 5;16(6):e146. doi: 10.2196/jmir.3077. PMID 24905070
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Vries Hd, Mesters I, van de Steeg H, Honing C. The general public's information needs and perceptions regarding hereditary cancer: an application of the Integrated Change Model. Patient Educ Couns. 2005 Feb;56(2):154-65. doi: 10.1016/j.pec.2004.01.002. PMID 15653244
- [Derived] Jimenez-Diaz A, Pierantonelli M, Morte Coscolin P, Salinas-Uhalte A, Quer-Palomas S, Rivera-Romero O, Herrero R, Fernandez-Luque L, Banos R, Berrios RC, de Arriba A. Digital Health Program to Support Family Caregivers of Children Undergoing Growth Hormone Therapy: Qualitative Feasibility Study. JMIR Pediatr Parent. 2025 Feb 5;8:e55023. doi: 10.2196/55023. PMID 39908086
- [Derived] Cervera-Torres S, Nunez-Benjumea FJ, de Arriba Munoz A, Chicchi Giglioli IA, Fernandez-Luque L. Digital health for emotional and self-management support of caregivers of children receiving growth hormone treatment: a feasibility study protocol. BMC Med Inform Decis Mak. 2022 Aug 13;22(1):215. doi: 10.1186/s12911-022-01935-1. PMID 35964116
- [Derived] Nunez-Benjumea FJ, Munoz AA, Callau MV, Fernandez-Luque L. Description of a Digital Health Platform for Emotional and Self-Management Support of Caregivers of Children Receiving Growth Hormone Treatment. Stud Health Technol Inform. 2022 Jan 14;289:290-292. doi: 10.3233/SHTI210916. PMID 35062149